CLINICAL TRIAL: NCT00028847
Title: A Dose-ranging Phase I/II Study of STI571 in Combination With Cytarabin in Patients With First Chronic Phase Chronic Myeloid Leukemia
Brief Title: Imatinib Mesylate and Cytarabine in Treating Patients With Newly Diagnosed Chronic Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Commissie Voor Klinisch Toegepast Onderzoek (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069141; CKTO-2001-03; HOVON-51CML; EU-20132; HOVON-CKTO-2001-03; NOVARTIS-CST1571ANL01
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2011-08

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cytarabine; Imatinib Mesylate

INTERVENTIONS:
Drug: cytarabine
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining imatinib mesylate and chemotherapy may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of imatinib mesylate plus cytarabine in treating patients who have newly diagnosed chronic myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of imatinib mesylate and cytarabine in patients with newly diagnosed chronic phase chronic myeloid leukemia.
* Determine the feasibility of this regimen as defined by dose-limiting toxicity of this regimen and treatment-related mortality in no more than 5% of these patients.
* Determine the rate and duration of molecular response, complete hematological response, and complete cytogenetic response in patients treated with this regimen.
* Determine the time to treatment failure of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of imatinib mesylate and cytarabine.

Patients receive oral imatinib mesylate alone once daily on days 1-21. Patients then receive oral imatinib mesylate once daily and cytarabine IV over 1-3 hours on days 1-7. Combination therapy repeats every 28-42 days for 2 courses. Patients then receive maintenance oral imatinib mesylate once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 5-20 patients receive escalating doses of imatinib mesylate and cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 5/5, 5/10, or 5/20 patients experience dose-limiting toxicity.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 30-60 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed chronic myeloid leukemia in first chronic phase (within the past 6 months)

  * Philadelphia-chromosome positive OR
  * bcr-abl rearrangement
* No prior treatment within the past 6 months other than hydroxyurea

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No hepatic dysfunction
* Bilirubin less than 2 times normal
* ALT less than 4 times normal

Renal:

* No renal dysfunction
* Creatinine less than 2.3 mg/dL

Cardiovascular:

* No severe cardiac dysfunction
* No New York Heart Association class II-IV heart disease

Pulmonary:

* No severe pulmonary disease

Other:

* HIV negative
* No severe neurologic disease
* No active uncontrolled infection
* No other active malignancy within the past 5 years except basal cell skin cancer or stage 0 cervical cancer
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent allogeneic transplantation with an HLA-A, B, DR-matched sibling donor or matched-unrelated donor

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No concurrent grapefruit or grapefruit juice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-04

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity and treatment-related toxicity per dose level

SECONDARY OUTCOMES:
Rate and duration of molecular response
Rate and duration of complete hematological response
Rate and duration of complete cytogenetic response
Time to treatment failure
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Cornelissen, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (16):
- Belgium (5):
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- Netherlands (11):
  - Meander Medisch Centrum, Amersfoort
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken - locatie Sophia, Zwolle

REFERENCES:
- [Result] Deenik W, Janssen JJ, van der Holt B, Verhoef GE, Smit WM, Kersten MJ, Daenen SM, Verdonck LF, Ferrant A, Schattenberg AV, Sonneveld P, van Marwijk Kooy M, Wittebol S, Willemze R, Wijermans PW, Beverloo HB, Lowenberg B, Valk PJ, Ossenkoppele GJ, Cornelissen JJ. Efficacy of escalated imatinib combined with cytarabine in newly diagnosed patients with chronic myeloid leukemia. Haematologica. 2010 Jun;95(6):914-21. doi: 10.3324/haematol.2009.016766. Epub 2009 Dec 16. PMID 20015886
- [Result] Deenik W, van der Holt B, Verhoef GE, Smit WM, Kersten MJ, Kluin-Nelemans HC, Verdonck LF, Ferrant A, Schattenberg AV, Janssen JJ, Sonneveld P, van Marwijk Kooy M, Wittebol S, Willemze R, Wijermans PW, Westveer PH, Beverloo HB, Valk P, Lowenberg B, Ossenkoppele GJ, Cornelissen JJ. Dose-finding study of imatinib in combination with intravenous cytarabine: feasibility in newly diagnosed patients with chronic myeloid leukemia. Blood. 2008 Mar 1;111(5):2581-8. doi: 10.1182/blood-2007-08-107482. Epub 2008 Jan 2. PMID 18172005
- [Derived] Thielen N, van der Holt B, Cornelissen JJ, Verhoef GE, Gussinklo T, Biemond BJ, Daenen SM, Deenik W, van Marwijk Kooy R, Petersen E, Smit WM, Valk PJ, Ossenkoppele GJ, Janssen JJ. Imatinib discontinuation in chronic phase myeloid leukaemia patients in sustained complete molecular response: a randomised trial of the Dutch-Belgian Cooperative Trial for Haemato-Oncology (HOVON). Eur J Cancer. 2013 Oct;49(15):3242-6. doi: 10.1016/j.ejca.2013.06.018. Epub 2013 Jul 19. PMID 23876833